CLINICAL TRIAL: NCT01484314
Title: A Phase II Study of Eltrombopag for the Treatment of Thrombocytopenia in Patients Undergoing Therapy for Relapsed Multiple Myeloma
Brief Title: Eltrombopag for Thrombocytopenia in Patients With Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nancy Berliner, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-373
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Thrombocytopenia; Multiple Myeloma
Keywords: Relapsed
MeSH Terms: conditions — Thrombocytopenia; Multiple Myeloma; Recurrence | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Migration Arm (Experimental): Administration of eltrombopag to support platelets during chemotherapy
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — 100mg (patients of East Asian descent will receive a dose of 50mg) orally dosed once daily starting 6 days prior to initiation of chemotherapy for a total of 11 days of treatment during two consecutive cycles of chemotherapy

SUMMARY:
Eltrombopag is a compound that may help stimulate the production of platelets. This drug has been used in treatment of low platelet counts caused by a disorder called idiopathic thrombocytopenic purpura and information from those other research studies suggests that Eltrombopag may help to maintain platelet counts in patients with relapsed multiple myeloma in this research study.

In this research study,the investigators are trying to determine if Eltrombopag is effective in maintaining platelet counts in patients who are being treated for relapsed multiple myeloma.

DETAILED DESCRIPTION:
You will take eltrombopag during two consecutive cycles of chemotherapy. During these two cycles you will be asked to complete the following for the research study in addition to any clinical exams or procedures that your regular doctor may order:

Study Drug(s): If you take part in this research study, you will be given a study drug-dosing calendar for each treatment cycle. Each treatment cycle lasts 27 days during which time you will be taking the study drug for 11 days on days 1 through 11.

Clinical Exams: You will have a physical exam on days 1, 11, and 21 of both cycles. You will be asked questions about your general health and specific questions about any problems that you might be having and any medications you may be taking. Your vital signs will be collected during this exam.

Performance status: Your ability to perform daily tasks will be assessed on days 1 and 27 of both cycles.

Blood Tests: You will have tests to check for safety performed on days 1, 7, 11, 20, and 27 of both cycles. You will have approximately 1-2 teaspoons of blood collected.

Concurrent Medications: Any changes to your medications will be recorded. Adverse Events: You be continually monitored for any changes to you health or well-being while you are on this study.

You will complete all subsequent cycles of chemotherapy procedures per standard of care for DFCI. During the subsequent cycles, you will not take eltrombopag.

After the final dose of the study drug: On Day 1 of cycle 3 of chemotherapy, you will complete the end of study/off study evaluations. The following procedures will be completed:

* Physical Exam, including vitals signs
* Performance status, which evaluates how you are able to carry on with your usual activities.
* Tumor Measurements: We will assess your tumor by blood tests and/or bone marrow aspirate and biopsy. If clinically indicated, you may have CT scans, bone scans or skeletal surveys
* Blood tests, routine tests to check for safety
* Concurrent Medications: Any changes to your medications will be recorded.

Follow-up:

We would also like to keep track of your medical condition for thirty days after your last dose of study drug. We would like to do this by having you return to have your blood counts checked once a week for 4 weeks and by calling you to check your condition and any changes to your health or well-being that may have occurred since you last took the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed multiple myeloma that is relapsed or refractory
* Patients may have had 1 or more prior chemotherapy regimens for multiple myeloma but none within the preceding 14 days
* Performance status (ECOG) ≤ 2
* Not pregnant or breastfeeding

Exclusion Criteria:

* Participants with a history of rapidly progressive disease [increase in tumor size (≥ 50%) as defined by standard myeloma markers ], pelvic irradiation, chemotherapy or radiotherapy within the preceding 14 days
* Participants may not be receiving any other study agents within 21 days prior to entry on the study.
* The use of growth factors other than erythropoiesis stimulating agents or G-CSF (Neupogen or Neulasta) during the study period.
* Participants with evidence of active thromboembolic disease or a history of thromboembolism within the preceding 6 months (excluding thrombosis of a central line).
* Participants with a documented history of genetic predisposition for thrombosis (anti-phospholipid antibody syndrome, AT-III deficiency, etc.), platelet disorder or bleeding disorder.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Individuals with a history of other malignancies are eligible only if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the preceding 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Berliner, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Migration Arm
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Migration Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants] — Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Region of Enrollment [Number; unit: participants] — Population: Terminated with 1 patient enrolled; no data due to patient privacy.

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of Platelet Count
Description: To determine the proportion of patients with relapsed multiple myeloma in whom eltrombopag maintains platelet counts at > 90% of baseline platelet counts with no more than 4 units of platelet transfusions at day 1 of Cycle 3 of chemotherapy
Time Frame: 2 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Migration Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Safety and Tolerability
Description: To determine whether eltrombopag administration results in an increased number of participants with adverse events.
Time Frame: 2 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Migration Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Grade 3/4 Thrombocytopenic Events
Description: To assess whether eltrombopag decreases the incidence of grade 3/4 thrombocytopenic events by day 1 of Cycle 3 of chemotherapy
Time Frame: 2 years
Population: Terminated with 1 patient enrolled; no data due to patient privacy.
Arm/Group | Migration Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AE assessment was ongoing from the start of study drug and up to day 30 post-treatment. Due to privacy concerns with enrollment of one patient, no data is provided.
Arm/Group | Migration Arm
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study is limited because it terminated early with only 1 patient enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No